CLINICAL TRIAL: NCT05613777
Title: The Effect of Multiple Doses of BI 425809 on the Pharmacokinetics of Multiple Doses of a Combination of Ethinylestradiol and Levonorgestrel Following Oral Administration in Healthy Premenopausal Female Subjects (an Open-label, Two-period, Fixed Sequence Design Trial With run-in Period)
Brief Title: A Study in Healthy Women to Test Whether BI 425809 Influences the Amount of a Contraceptive in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0036; 2022-500050-42-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination; BI 425809

STUDY DESIGN:
Intervention Model Description: Fixed sequence: Run in period-Reference-Treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microgynon®(Run-in)/Microgynon® (treatment reference, R)/ Microgynon®+BI 425809 (treatment test, T) (Experimental)
  Interventions: Drug: Microgynon®; Drug: BI 425809

INTERVENTIONS:
Drug: Microgynon® — ethinylestradiol (EE) and levonorgestrel (LNG)
Drug: BI 425809 — BI 425809

SUMMARY:
The main objective of this trial is to investigate the possible effect of multiple oral doses of BI 425809 on the steady state pharmacokinetics of ethinylestradiol (EE) and levonogestrel (LNG) (administered as the combined oral contraceptive Microgynon®).

ELIGIBILITY:
Inclusion Criteria:

* Healthy premenopausal female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure(BP), Pulse rate (PR)), 12-lead Electrocardiogram (12-lead ECG), and clinical laboratory tests without any clinically significant abnormalities.
* Age of 18 to 35 years (inclusive).
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive).
* Signed and dated written informed consent in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Female subjects who meet any of the following criteria starting from at least 30 days before the first administration of BI 425809 and until 30 days after trial completion:

  * Use of adequate contraception, e.g. non-hormonal intrauterine device plus condom.
  * Sexually abstinent.
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment).
  * Surgically sterilised (including hysterectomy).

Exclusion Criteria:

Subjects will not be allowed to participate, if any of the following general criteria apply:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm).
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair).
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders.
* History of relevant orthostatic hypotension, fainting spells, or blackouts. Further exclusion criteria apply.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss ) | Up to 22 days
Maximum measured concentration of the analyte in plasma at steady state over (Cmax,ss) | Up to 22 days
Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ(Cmin,ss) | Up to 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Madari S, Balavarca Y, Shatillo Y, Reuteman-Fowler C, Desch M. The Effect of Multiple Oral Doses of a Glycine Transporter 1 Inhibitor, Iclepertin (BI 425809), on the Steady-state Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinylestradiol and Levonorgestrel: a Phase I Clinical Trial in Healthy Females. Clin Drug Investig. 2025 Oct;45(10):767-779. doi: 10.1007/s40261-025-01472-5. Epub 2025 Sep 4. PMID 40906309
- See also: Related Info — https://www.mystudywindow.com